CLINICAL TRIAL: NCT02427386
Title: Phase 4 Randomized Controlled Trial of Dynamized Estrogen in Individualized Homeopathic Treatment of Chronic Pelvic Pain of Endometriosis
Brief Title: Homeopathic Treatment of Chronic Pelvic Pain in Women With Endometriosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcus Zulian Teixeira, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMUSP
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Endometriosis; Pelvic pain; Homeopathy; RCT
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dynamized estrogen in alcohol solution (Active Comparator): Dynamized estrogen (17-beta estradiol) in the 12cH, 24cH and 18cH potencies.
  Interventions: Drug: dynamized estrogen
- placebo (alcohol solution) (Placebo Comparator): This arm received alcohol solution during the 24-week study duration.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dynamized estrogen — The dosage of the homeopathic medicine or placebo will be of 3 drops, 2 times a day throughout the period of study, and can be reduced in case of finding of homeopathic aggravation of symptoms. 30 ml bottles will be sufficient for the proposed dosage every 8 weeks of treatment (bimensal period).
  Other Names: dynamized 17-beta estradiol
  Arms: dynamized estrogen in alcohol solution
Drug: placebo — The dosage of the placebo (alcohol solution) will be of 3 drops, 2 times a day throughout the period of study.
  Other Names: alcohol solution
  Arms: placebo (alcohol solution)

SUMMARY:
Endometriosis is a chronic inflammatory disease that causes pelvic pain difficult to treat. In view of this, many patients seek assistance in complementary and alternative medicine, including homeopathic treatment. The absence of evidence in the literature raises controversy about the effectiveness of homeopathic treatment in endometriosis. The aim of this randomized trial is to evaluate the effectiveness of dynamized estrogen compared to placebo in the treatment of chronic pelvic pain of endometriosis.

DETAILED DESCRIPTION:
This is a randomized, double-blind and placebo controlled trial using individualised homeopathic medicine (dynamized estrogen) to treat chronic pelvic pain of endometriosis. Patients with endometriosis, chronic pelvic pain and a set of signs and symptoms similar to those of the estrogen adverse events will be recruited in the Sector of Endometriosis of the Clinical Division of Gynaecological of the Hospital das Clínicas of the Faculty of Medicine of the University of Sao Paulo. The selection process was carried out through the analysis of medical charts and self-completing of structured questionnaires. Satisfied the inclusion criteria, fifty patients were randomly and distributed to receive dynamized estrogen or placebo. The primary clinical outcome is the severity of the chronic pelvic pain. Statistical analysis will be by intention-to-treat and per protocol comparing homeopathic drug with placebo after 24 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

primary inclusion criteria:

* aged between 18 and 45;
* diagnosis of endometriosis (endometrial ectopia) confirmed by imaging test (MRI or TVUS) or laparoscopy (biopsy);
* chronic pelvic pain refractory to conventional hormone treatments and with intensity ≥ 5 on the visual analog pain scale (VAS-Pain: 0-10 points);

secondary inclusion criteria:

* symptomatic individualization of patients according to adverse events of estrogen (minimum syndrome of maximum value).

Exclusion Criteria:

* absence of clinical and laboratory diagnosis of menopause or
* premature ovarian failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
chronic pelvic pain (measured by visual analog scale (VAS-Pain) | 24 weeks (6 months)
  chronic pelvic pain (dysmenorrhoea, dyspareunia, acyclic pelvic pain depth, cyclic intestinal change and cyclic urinary change) measured by visual analog scale (VAS-Pain)

SECONDARY OUTCOMES:
36-Item Short-Form Health Survey (SF-36) | 24 weeks (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Z Teixeira, PhD, Principal Investigator — University of Sao Paulo General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teixeira MZ. 'New Homeopathic Medicines' database: A project to employ conventional drugs according to the homeopathic method of treatment. European Journal of Integrative Medicine 5(3): 270-278, 2013.
- [Background] Teixeira MZ, Podgaec S, Baracat EC. Protocol of randomized controlled trial of potentized estrogen in homeopathic treatment of chronic pelvic pain associated with endometriosis. Homeopathy. 2016 Aug;105(3):240-249. doi: 10.1016/j.homp.2016.03.002. Epub 2016 May 13. PMID 27473545
- [Background] Teixeira MZ, Podgaec S, Baracat EC. Potentized estrogen in homeopathic treatment of endometriosis-associated pelvic pain: A 24-week, randomized, double-blind, placebo-controlled study. Eur J Obstet Gynecol Reprod Biol. 2017 Apr;211:48-55. doi: 10.1016/j.ejogrb.2017.01.052. Epub 2017 Jan 25. PMID 28187404
- [Result] Teixeira MZ. Homeopathic use of modern medicines: utilisation of the curative rebound effect. Med Hypotheses. 2003 Feb;60(2):276-83. doi: 10.1016/s0306-9877(02)00386-9. PMID 12606247
- [Result] Teixeira MZ. New homeopathic medicines: use of modern drugs according to the principle of similitude. Homeopathy. 2011 Oct;100(4):244-52. doi: 10.1016/j.homp.2011.01.002. PMID 21962199
- See also: New homeopathic medicines: use of modern drugs according to the principle of similitude — http://www.newhomeopathicmedicines.com